CLINICAL TRIAL: NCT03023878
Title: 20150288 A Phase 2 Open-label Study Investigating the Safety and Efficacy of Blinatumomab After Frontline R-Chemotherapy in Adult Subjects With Newly Diagnosed High-risk Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Safety and Efficacy of Blinatumomab in Adults With Newly Diagnosed High-risk Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150288; 2016-002190-35 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2017-01-18 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: High-risk Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — blinatumomab; Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Blinatumomab was administered as a continuous intravenous (IV) infusion. Cycle 1 was 12 weeks (84 days) in duration with step dosing of 9 µg/day for 7 days, 28 µg/day for 7 days, 112 µg/day for 6 weeks, followed by a 4-week treatment free time.
  An optional 4-week Cycle 2 of blinatumomab was available for participants whose disease did not progress, with step dosing of 9 µg/day for 7 days, 28 µg/day for 7 days, and 112 µg/day for 14 days.
  There was a safety follow-up for 30 days. And a long-term follow-up of up to 8 months for a maximum of 1 year from first dose of blinatumomab or until participant death.
  Interventions: Drug: Blinatumomab; Drug: Investigator's Choice Chemotherapy; Drug: Dexamethasone

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab monotherapy was supplied in single-use sterile glass injection vials and administered as an IV infusion.
  Other Names: AMG103; BlinCyto
Drug: Investigator's Choice Chemotherapy — During the run-in period participants received 6 cycles of standard of care rituximab-chemotherapy dosed per investigator's institution standard as follows:
  * R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine,prednisone)
  * R-DA-EPOCH (rituximab and dose adjusted-etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin) or
  * R-CHOEP (rituximab and cyclophosphamide, doxorubicin, vincristine, prednisone, and etoposide).
Drug: Dexamethasone — Dexamethasone 20 mg IV: within 1 hour prior to start of treatment in each treatment cycle, and within 1 hour prior to dose-step (increase).
  Other Names: corticosteroid

SUMMARY:
A phase 2, multicenter, open-label, single arm clinical trial in adults with newly diagnosed aggressive high-risk DLBCL.

DETAILED DESCRIPTION:
The safety profile of blinatumomab after frontline rituximab (R)-chemotherapy, consisting of either R-CHOP (14 or 21) (rituximab/cyclophosphamide/doxorubicin/vincristine/prednisone) or R-DA-EPOCH (rituximab and dose adjusted-etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin), or R-CHOEP (rituximab and cyclophosphamide, doxorubicin, vincristine, prednisone, and etoposide), will be determined. The study will consist of a screening period of up to 14 days, a standard of care (SOC) R-chemotherapy run-in period of approximately 21 weeks, a 12 to 16 week blinatumomab treatment period, a 30-day safety follow-up visit, and a long-term follow-up period that begins after the safety follow-up visit is completed until 1 year from the first dose blinatumomab.

ELIGIBILITY:
Inclusion criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age ≥ 18 at time of informed consent
* Subject must have untreated histologically proven high-risk DLBCL defined by atleast one of the following:

  * International Prognostic Index (IPI) for Diffuse Large B-cell Lymphoma 3 to 5 (representing high intermedidate - high ratings),
  * Double-hit or higher or double protein expression
* Eastern Cooperative Oncology Group performance status ≤ 2.
* Subject meets the criteria per investigator's institution to receive standard of care (SOC) rituximab-chemotherapy (ie, R-CHOP [14 or 21] or R-DA-EPOCH or R-CHOEP) of 6 cycles. Subjects may be enrolled on study prior to cycle 1 or cycle 2 of SOC R-chemotherapy
* Adequate organ and bone marrow function determined within 14 days prior to enrollment defined as:

  * Hematological: Absolute neutrophil count ≥1*10^9/L; Platelet count ≥75*10^9/L;Hemoglobin ≥8g/dL
  * Renal: Creatinine clearance ≥50mL/min;
  * Hepatic: Aspartate aminotransferase/Alanine aminotransferase <3*upper limit of normal (ULN); Total bilirubin <2*ULN (unless Gilbert's Disease or if liver involvement with lymphoma)
* Subject must have completed 6 cycles of SOC R-chemotherapy and achieved CR, PR or stable disease by PET/CT performed 3 weeks (± 3 days) after cycle 6 of SOC R-chemotherapy. Subjects with progressive disease (PD) are not eligible for treatment with blinatumomab and will end the study.

Exclusion Criteria:

* Clinically relevant central nervous system (CNS) pathology requiring treatment such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, and psychosis
* Evidence of CNS involvement with DLBCL at disease evaluation obtained prior to starting blinatumomab
* Current autoimmune disease or history of autoimmune disease with potential of CNS involvement
* Subject has active infection requiring systemic therapy
* Prior anti-CD19 therapies
* Known infection with HIV or chronic infection with hepatitis B virus or hepatitis C virus
* History of other malignancy within the past 3 years with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ
* Subject has known hypersensitivity to immunoglobulins or any of the products or components to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge.
* History/evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed while receiving blinatumomab and for an additional 48 hours after the last treatment dose of blinatumomab.
* Currently receiving treatment in another investigational device or drug study or less than 30 days since ending treatment on another investigational device or drug study. Other investigational procedures while participating in this study are excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (24):
- United States (8):
  - Research Site, Chicago, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, New Brunswick, New Jersey
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
- France (2):
  - Research Site, Créteil
  - Research Site, Paris
- Germany (2):
  - Research Site, Dresden
  - Research Site, Ulm
- Spain (7):
  - Research Site, Seville, Andalusia
  - Research Site, Salamanca, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, Bristol
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Katz DA, Morris JD, Chu MP, David KA, Thieblemont C, Morley NJ, Khan SS, Viardot A, Martin Garcia-Sancho A, Rodriguez-Garcia G, Bastos-Oreiro M, Lee ST, Kormany W, Chen Y, Wong HL, Anderson AA, Katlinskaya Y, Avilion AA, Dai T, Gonzalez-Barca E. Open-label, phase 2 study of blinatumomab after frontline R-chemotherapy in adults with newly diagnosed, high-risk DLBCL. Leuk Lymphoma. 2022 Sep;63(9):2063-2073. doi: 10.1080/10428194.2022.2064981. Epub 2022 May 3. PMID 35503708
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 centers in the European Union (France, Germany, Spain, and the United Kingdom), the United States, and Canada.
  Of the 54 subjects screened, 47 subjects were enrolled.
Pre-assignment Details: The study consisted of a standard of care rituximab-chemotherapy Run-in Period of approximately 21 weeks, a 12- to 16-week blinatumomab Treatment Period, a 30-day safety follow-up, and a Long-term Follow-up Period up to 1 year from the first dose of blinatumomab, or until participant death, whichever occurred first.
Period: Pre-Study Run-In Period
Arm/Group | Blinatumomab
Started (Standard of Care (SOC) rituximab (R)-chemotherapy Analysis Set.) | 47
Completed | 30
Not Completed | 17
Not completed — Protocol-specified criteria | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 5
Period: Between Run-In and Treatment Periods
Arm/Group | Blinatumomab
Started | 30
Completed | 28
Not Completed | 2
Not completed — Protocol-specified criteria | 2
Period: Treatment Period
Arm/Group | Blinatumomab
Started | 28
Started Cycle 1 (Full analysis set (FAS)) | 28
Started Cycle 2 | 11
Completed | 25
Not Completed | 3
Not completed — Disease Progression | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Period: Long Term Follow-Up Period
Arm/Group | Blinatumomab
Started (Treatment period participants are followed) | 28
Completed | 26
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least 1 dose of blinatumomab.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.1)
Age, Customized [Count of Participants; unit: Participants] — Note the overlapping age groups
  Participants
    < 65 years | 18
    >=65 years | 10
    <75 years | 25
    >=75 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black and African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 21
  Other | 4
Disease Stage at Time of Diagnosis [Count of Participants; unit: Participants] — * Stage I - Only one lymph node region is involved, only one lymph structure is involve
  * Stage IE - Only one extranodal site (IE) is involved.
  * Stage II - Two or more lymph node regions or lymph node structures on the same side of the diaphragm are involved.
  * Stage III - Lymph node regions or structures on both sides of the diaphragm are involved.
  * Stage IV - There is widespread involvement of a number of organs or tissues other than lymph node regions or structures, such as the liver, lung, or bone marrow.
  Participants
    Stage I | 0
    Stage IE | 1
    Stage II | 0
    Stage III | 5
    Stage IV | 22
International Prognostic Index Score at Diagnosis [Count of Participants; unit: Participants] — IPI score is an aid in predicting the prognosis of patients
  * Low risk (0-1 points) - 5-year survival of 73%
  * Low-intermediate risk (2 points) - 5-year survival of 51%
  * High-intermediate risk (3 points) - 5-year survival of 43%
  * High risk (4-5 points) - 5-year survival of 26%
  Participants
    Score 2 | 2
    Score 3 | 17
    Score 4 | 7
    Score 5 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent (Blinatumomab) Adverse Events
Description: Overall incidence and severity of treatment-emergent adverse events occurring during the blinatumomab investigative product (IP) treatment period graded by investigators according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and based on the scale:
  Grade 1 = Mild - transient or mild discomfort; Grade 2 = Moderate - mild to moderate limitation in activity, assistance may be needed; minimal medical intervention required; Grade 3 = Severe - marked limitation in activity, assistance usually required; medical intervention required, hospitalization is possible; Grade 4 = Life threatening - extreme limitation in activity, assistance required; medical intervention, hospitalization or hospice care probable; Grade 5 = death.
Time Frame: From the start of first infusion of IP to 30 days after the end of last infusion of IP; median (min, max) treatment duration was 56 (16, 84) days
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
Participants
  TEAE | 28
  TEAE severity grade >=3 | 11
  TEAE severity grade >=4 | 5
  Serious TEAE | 7
  TEAE leading to interruption of IP | 3
  Serious TEAE leading to interruption of IP | 2
  TEAE leading to discontinuation of IP | 2
  Serious TEAE leading to discontinuation of IP | 1
  Fatal TEAEs | 0

2. Primary Outcome: Participants With Treatment-Emergent Adverse Events Related to Blinatumomab Treatment
Description: Overall incidence and severity of treatment-emergent adverse events deemed by investigators to be related to blinatumomab treatment. Severity was graded by investigators according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and based on the scale:
  Grade 1 = Mild - transient or mild discomfort; Grade 2 = Moderate - mild to moderate limitation in activity, assistance may be needed; minimal medical intervention required; Grade 3 = Severe - marked limitation in activity, assistance usually required; medical intervention required, hospitalization is possible; Grade 4 = Life threatening - extreme limitation in activity, assistance required; medical intervention, hospitalization or hospice care probable; Grade 5 = death.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
Participants
  Treatment-related TEAE | 23
  Related TEAE severity grade >=3 | 9
  Related TEAE severity grade >=4 | 3
  Related Serious TEAE | 5
  Related TEAE leading to interruption of IP | 3
  Related Serious TEAE leading to interruption of IP | 2
  Related TEAE leading to discontinuation of IP | 2
  Related Serious TEAE leading to discon of IP | 1
  Related and Fatal TEAEs | 0

3. Secondary Outcome: Overall Objective Response Rate (ORR) Expressed as the Percentage of Participants Achieving Complete Metabolic Response (CMR) and Partial Metabolic Response (PMR) Using Lugano 2014 Criteria During Cycle 1 and During Treatment Period
Description: Tumor response assessment was performed by a central reader according to modified Lugano classification using PET/CT scan. Overall objective response rate (ORR) is the percentage of participants with a best overall response of complete metabolic response (CMR) or partial metabolic response (PMR). CMR: a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with/without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PMR: a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline.
Time Frame: Cycle 1: Day 78 (3 weeks following end of Cycle 1 IP treatment) Treatment Period: Either the Cycle 1 timeframe or approximately Day 128 (3 weeks after Cycle 2 ended) for participants who completed Cycle 2
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
percentage of participants
  Cycle 1 | 89.3 [71.8 to 97.7]
  Entire Treatment Period | 92.9 [76.5 to 99.1]

4. Secondary Outcome: Kaplan-Meier Estimates for Duration of Response
Description: Duration of response was calculated only for responders during cycle 1. For participants who had CR or PR on the PET/CT scan at the end of the run-in period, response was measured from the start of blinatumomab treatment. For participants who had stable disease at the end of the run-in period, duration was calculated from documentation of the first assessment of either PR or CR on blinatumomab.
  Progression was defined as the first diagnosis of progressive metabolic response/progressive disease based on PET/CT scan per central or investigator review during the treatment period or relapse based on clinical tumor assessment during the long-term follow up period.
  Response duration was calculated until the start of new anti-tumor treatment (excluding any stem cell transplantation), PD, or death, whichever was the earliest event. Participants who did not have new anti-tumor treatment (excluding stem cell transplantation), PD, or death were censored at the last tumor assessment date.
Time Frame: The median (range) follow-up time was 11.5 (8.2, 14.5) months
Population: Responder Analysis Set includes all participants in the FAS that achieve objective response (CR or PR as per the Lugano classification) on the PET/CT scan.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
months | NA [NA to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Complete Response Rate Expressed as the Percentage of Participants Achieving Complete Metabolic Response (CMR) Using Lugano 2014 Criteria During Cycle 1 and During Treatment Period
Description: Tumor response assessment was performed by a central reader according to modified Lugano classification using PET/CT scan.
  CMR: a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with/without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology.
Time Frame: as for outcome 3
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
percentage of participants
  Cycle 1 | 85.7 [67.3 to 96.0]
  Entire Treatment Period | 89.3 [71.8 to 97.7]

6. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS) From First Dose of Blinatumomab
Description: OS was calculated as the time from the date of first IP infusion until death due to any cause. Participants who are alive at the date that triggers the analysis were censored at the date last known to be alive.
  Months were calculated as days from the first dose date of blinatumomab to death/censor date, divided by 30.5.
Time Frame: The median (range) follow-up time was 12.0 (10.7, 14.5) months.
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
months | NA [NA to NA] — Could not be estimated due to the low number of events

7. Secondary Outcome: Kaplan-Meier Estimates for Progression Free Survival (PFS) From First Dose of Blinatumomab
Description: PFS was calculated as the time from the date of first IP infusion until the date of diagnosis of progression of DLBCL or the date of death, whichever was the earliest. The diagnosis of progression of DLBCL was defined as the first diagnosis of progressive metabolic response/progressive disease based on PET/CT scan per central or investigator review during the treatment period or relapse based on clinical tumor assessment during the long-term follow up period. Participants who were alive and did not have progression were censored at the last evaluable non-missing tumor assessment date prior to the analysis trigger date.
Time Frame: The median (range) follow-up time was 12.0 (8.2, 14.5)
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
months | NA [NA to NA] — Could not be estimated due to the low number of events

8. Secondary Outcome: Percentage of Participants Who Had Hematopoietic Stem Cell Transplantation (HSCT)
Description: Percentage of participants who had HSCT during the Long Term Follow-Up Period.
Time Frame: Day 1 up to 14.5 months
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
percentage of participants | 3.6 [0.1 to 18.3]

9. Secondary Outcome: Pharmacokinetics (PK) Results for Blinatumomab: Steady-State Concentrations at Week 1, Week 2 and Week 3 for Cycle 1
Description: The steady-state serum concentration (Css), summarized as the observed concentrations collected after at least 10 hours after the start of continuous IV infusion.
  PK blood samples were analyzed in a central lab.
Time Frame: Day 2 at least 24 hours after blinatumomab was started and on Day 9 and Day 16 at least 24 hours after blinatumomab dose was increased in the cycle
Population: Pharmacokinetic Analysis Set: participants who received any infusion of blinatumomab and had at least one PK sample collected
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
pg/mL
  Cycle 1 Week 1: 9 mcg/day: number analyzed (Participants) | 26
  Cycle 1 Week 1: 9 mcg/day | 288 (289)
  Cycle 1 Week 2: 28 mcg/day | 795 (280)
  Cycle 1 Week 3: 112 mcg/day: number analyzed (Participants) | 26
  Cycle 1 Week 3: 112 mcg/day | 3160 (782)

10. Secondary Outcome: Pharmacokinetics (PK) Results for Blinatumomab: Clearance for Cycle 1
Description: PK blood samples were analyzed in a central lab.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/Hour
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
L/Hour | 1.61 (0.496)

ADVERSE EVENTS:
Time Frame: Mortality is reported for all enrolled participants from enrollment in the Run-in Period to the end of long-term follow-up. Adverse events are reported from the first dose of blinatumomab through 30 days after last dose; median duration of treatment was 56 days. In addition, serious adverse events related to blinatumomab collected during the long-term follow-up period are reported; median time on follow-up was 12 months.
Description: All-cause mortality data are reported for all participants who enrolled in the Run-in Period. Adverse events are reported for all participants who received at least one dose of blinatumomab in the Treatment Period. During the long-term follow-up period, only serious adverse events related to blinatumomab were collected.
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 3/47
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=28)
Neutropenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 2
Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Aphasia (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=28)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chills (General disorders) | 3
Fatigue (General disorders) | 8
Pyrexia (General disorders) | 10
Cytokine release syndrome (Immune system disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Ataxia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 9
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03023878/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03023878/SAP_001.pdf